CLINICAL TRIAL: NCT05449275
Title: The Effects Of Faradic Current Versus Ankle-Foot Orthosis In Patients With Foot Drop Due To Stroke
Brief Title: Effects Of Faradic Current Versus Ankle-Foot Orthosis In Patients With Foot Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-FSD-00264
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Foot Drop
Keywords: Stroke; Faradic Current; Ankle-Foot Orthosis; Foot Drop; Randomized Control Trial
MeSH Terms: conditions — Peroneal Neuropathies; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faradic current (Experimental): This study will use the faradic current for treating foot drop. In Group A 15 number of patient with foot drop will get the 40 minutes of session with the frequency of 50-100hz alternative three days / week for 25 weeks
  Interventions: Other: Faradic current
- Ankle foot orthosis (Experimental): Group B will get the treatment by Ankle foot orthosis.In group B 15 patients with foot drop will get the session alternative three days/week for 25 weeks. All participants have to use Ankle foot orthosis on a daily basis and patients have to walk for 10 minutes without walking aid.
  Interventions: Other: Ankle foot orthosis

INTERVENTIONS:
Other: Faradic current — The most common Electrical stimulation applied for foot drop is faradic current. Faradic current provides the strength and improvement to volitational muscles and increase the coordination and reduce spasticity.
  Arms: Faradic current
Other: Ankle foot orthosis — AFO is most commonly used technique but it also has some disadvantage mainly is the movement in limited direction and also in development of contractures and may have the problem in standing from chair
  Arms: Ankle foot orthosis

SUMMARY:
This research aims to compare changes in gait quality and function between faradic current & Ankle foot orthosis with stroke related foot drop

DETAILED DESCRIPTION:
Randomized control trial study will be carried out at different health care units when synopsis will be approved. Enrollment of patients will be done by using purposive sampling technique. The selection of the patients will be done on the basis of exclusion criteria and inclusion criteria. The patients enrolled will be divided into 2 groups. Group A patients will be given faradic current on the other hand group B patients will be provided with ankle foot orthosis. The assessment of the patient will be done after 6 months and the outcome tools used will be 10-meter walk test, stroke impact scale, 6-meter walk test, Berg balance scale, Time up and go test. The data of the patient will be noted before giving treatment and after treatment and will be compared after 6 months. Consent will be taken from each patient. Statistical Package of Social Sciences Version 20 will be used for the entry and analysis of data

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been affected by stroke
* Good communication skills so the patient can follow the instructions
* Patients of both genders with any age group

Exclusion Criteria:

* Impairment in lower limb other that foot drop
* Patient suffering with any cardiovascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 12th Week
  The Berg Balance Scale is used to objectively determine a patient's ability or inability to safely balance during a series of predetermined tasks.
Stroke impact scale | 12th Week
  The Stroke Impact Scale assesses other dimensions of health related quality of life: emotion, communication, memory and thinking, and social role function. *The first four of these domains may be combined into one physical domain, but the others must be scored separately.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No